CLINICAL TRIAL: NCT03116997
Title: Randomized Controlled Assessor Blinded Clinical Trial of Sugammadex Versus Neostigmine /Glycopyrrolate for Reversal of Rocuronium Induced Neuromuscular Blockade: Time to Discharge From Post Anesthesia Care Unit and Patient Satisfaction With Recovery
Brief Title: Study of Recovery of Strength After Surgery Comparing Two Different Medications for Reversal of Muscle Relaxant
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-207
Record Dates: First submitted 2017-04-12; First posted 2017-04-17 (Actual); Results first posted 2023-03-07 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2023-02

CONDITIONS: Surgery
Keywords: neuromuscular blockade; sugammadex; SUG; neostigmine; NEO/GLYCO; 17-207
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Neuromuscular blockade reversed with neostigmine/gly (Experimental)
  Interventions: Drug: Neostigmine+glycopyrrolate
- Neuromuscular blockade reversed with sugammadex (Active Comparator)
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Neostigmine+glycopyrrolate — At the conclusion of surgery neuromuscular blockade reversed with neostigmine/glycopyrrolate
  Arms: Neuromuscular blockade reversed with neostigmine/gly
Drug: Sugammadex — At the conclusion of surgery neuromuscular blockade reversed with sugammadex
  Arms: Neuromuscular blockade reversed with sugammadex

SUMMARY:
The purpose of this study is to compare two different medications (neostigmine/glycopyrrolate and sugammadex) to see if one drug improves patient comfort regarding the return of muscle strength after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients age 18 years of age or greater who are capable of giving consent
* Undergoing surgical procedures of expected length 6 </= hours requiring NMB

Exclusion Criteria:

* Pregnancy
* History of documented anaphylaxis or contraindication to any of the study medications
* Active coronary disease with a positive cardiac stress test
* History of severe chronic obstructive pulmonary disease (COPD) defined as an FEV1 < 50% of predicted
* Serum Creatinine >/= 2.0 mg/dL
* Severe hepatic dysfunction accompanied by coagulopathy

  * Definition:
  * Known liver Disease AND
  * INR > 1.5 (except for patients on anticoagulants) AND
  * Platelet count <100,00/ul without other obvious cause
* Chronic sustained release opioid for > 2 weeks duration pre op (in the 30 days prior to surgery)
* Use of toremifene
* Significant cognitive impairment or documented psychologic impairment
* Myasthenia gravis or other neuromuscular disease
* Patients who are not eligible for standard anesthetic induction, eg, those needing rapid sequence induction or awake fiberoptic bronchial intubation.
* American Society of Anesthesiologists (ASA) Status > 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: German Echeverry, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Memoral Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memoral Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://mskcc.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Neuromuscular Blockade Reversed With Neostigmine/Gly | Neuromuscular Blockade Reversed With Sugammadex
Started | 100 | 101
Completed | 100 | 101
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neuromuscular Blockade Reversed With Neostigmine/Gly | Neuromuscular Blockade Reversed With Sugammadex | Total
Number analyzed (Participants) | 100 | 101 | 201
Age, Continuous [Median (Full Range); unit: years] | 55 [35 to 77] | 54 [21 to 83] | 55 [21 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 69 | 131
  Male | 38 | 32 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 13
  Not Hispanic or Latino | 94 | 94 | 188
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 7 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 11 | 20
  White | 86 | 73 | 159
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 10 | 14
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 100 | 101 | 201

OUTCOME MEASURES:

1. Primary Outcome: Measure Participants' Recovery Time Post-Surgery
Description: Determine whether SUG, as compared to NEO decreases time for patients to be ready for discharge from the PACU post-surgery.
Time Frame: 1 day
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Neuromuscular Blockade Reversed With Neostigmine/Gly | Neuromuscular Blockade Reversed With Sugammadex
Number analyzed (Participants) | 100 | 101
hours | 3.59 [2.49 to 5.09] | 3.62 [2.80 to 5.87]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Neuromuscular Blockade Reversed With Neostigmine/Gly | Neuromuscular Blockade Reversed With Sugammadex
All-Cause Mortality (participants affected / at risk) | 14/100 | 16/101
Serious Adverse Events (participants affected / at risk) | 2/100 | 2/101
Other Adverse Events (participants affected / at risk) | 0/100 | 0/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neuromuscular Blockade Reversed With Neostigmine/Gly (N=100) | Neuromuscular Blockade Reversed With Sugammadex (N=101)
Abdominal infection (Infections and infestations) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Kidney anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1
Pancreatic anastomotic leak (Injury, poisoning and procedural complications) | 0 | 2
Sepsis (Infections and infestations) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-17): https://cdn.clinicaltrials.gov/large-docs/97/NCT03116997/Prot_SAP_000.pdf